CLINICAL TRIAL: NCT04291118
Title: A Comparative Study Assessing Improvement in Cognitive Deficit Secondary to CRS in Patients Treated With Medical Vs Surgical Management: A Prospective Trial
Brief Title: Assessing Improvement in Cognitive Deficit in CRS in Patients Treated With Medical Vs Surgical Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Amin Javer, Clinical Professor, St. Paul's Hospital, Canada
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H19-03659
Record Dates: First submitted 2020-02-25; First posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Chronic Sinusitis
Keywords: Endoscopic Sinus Surgery; Medical Management; Cognitive Dysfunction; Modified Mini Mental State Examination
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Budesonide

STUDY DESIGN:
Intervention Model Description: New patients diagnosed with CRS (with or without polyps) who will receive medical or/and surgical management will be recruited for the study. They will be separated into one of 3 study arms based on the clinical care they require.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Medical Management and Sinus Surgery in private system (Other): These patients will first receive medical management for their symptoms and then will undergo sinus surgery much earlier than the other group as they will include patients being operated in the private system.
  Interventions: Procedure: Private system endoscopic sinus surgery
- Medical Management and Sinus Surgery in public system (Other): These patients will first receive medical management for their symptoms, and then will undergo sinus surgery after a waiting period of at least 1 year since they are on the public wait-list.
  Interventions: Procedure: Public system endoscopic sinus surgery
- Medical Management Only (Other): These patients will only receive medical management for their symptoms as they will not require sinus surgery.
  Interventions: Drug: Budesonide

INTERVENTIONS:
Procedure: Private system endoscopic sinus surgery — Patients that will undergo endoscopic sinus surgery though the private system. Beforehand they could of used medical management including, budesonide for their symptoms.
  Arms: Medical Management and Sinus Surgery in private system
Procedure: Public system endoscopic sinus surgery — Patients that undergo endoscopic sinus surgery though the public system after waiting for at least 1 year. Beforehand they could of used medical management, including budesonide for their symptoms.
  Arms: Medical Management and Sinus Surgery in public system
Drug: Budesonide — Patients will receive medical management for their symptoms that will consist of topical nasal steroid, budesonide and any other required medication for their disease.
  Arms: Medical Management Only

SUMMARY:
Chronic rhinosinusitis presents with a plethora of symptoms including non-rhinologic symptoms such as depression, sleep disturbances & the more recently recognized cognitive dysfunction. It has recently been identified that sinus specific treatments such as endoscopic sinus surgery can improve cognitive outcomes in patients with cognitive deficit secondary to chronic inflammation in the upper and lower airway. However, it remains to be seen whether or not offering surgery to these patients at an earlier date has an impact on the degree of improvement on cognitive function in comparison to patients who have to wait long periods for their treatment.

DETAILED DESCRIPTION:
Purpose To compare the improvement in cognitive deficit after medical management and surgical management in the treatment of Chronic Rhinosinusitis.

Hypothesis Cognitive deficit secondary to chronic rhinosinusitis will show a greater improvement with surgical management when compared to medical management.

Cognitive deficit secondary to chronic rhinosinusitis will improve quicker postoperatively for patients offered endoscopic sinus surgery earlier than for those who are placed on long waitlists for surgery

Study Design:

This is a prospective cohort series to be conducted at the St. Paul's Sinus Centre. All patients recruited into the study would have been diagnosed with chronic rhinosinusitis and will be subjected to appropriate and standardized medical management. They will be subjected to surgical management if they are not completely relieved of their symptoms. Prior to medical or surgical management, they will be subjected to the modified mini mental state examination to assess their baseline and post treatment (medical and surgical) cognitive function.

Data storage and safeguards The data will be stored on a password protected computer at St. Paul's Hospital in the Department of Otolaryngology on an encrypted Microsoft excel spreadsheet. The computer containing study data will be password-protected for access only by the principal investigator, co-investigator and study coordinator stored in a locked office, and backed-up remotely on to a secured hospital server. All hard copy documents will be kept in binders, in the Principal Investigator's office in a locked cabinet.

Patients participating in the study will all be assigned random study ID numbers. The study code is not derived from or related to the information about the individual, i.e., name, SIN, PHN, hospital number, DOB, address, or unique characteristic. These numbers will be used on all study documentation. Participant names are being stored separately from study data in a master list with the study ID numbers.

Data Monitoring Patients will continue to be assessed at routine follow up visits. Statistics will be completed after the study is complete on its objectives. Data will be also monitored on a continuous basis.

Statistical Analysis

Descriptive statistics will be used to summarize all demographic data, comorbidities, and adverse effects reported by the patients. Paired student t-tests will be applied to investigate the difference between the mean 3M Examination scores, MLK scores, SNOT-22 scores, before commencement of each treatment arm and subsequent MLK scores, SNOT-22 scores after treatment is complete. A running total of the treatment costs for each patient will be maintained. One way Anova test will be applied to investigate the difference between the mean costs for each treatment arm. Probability values less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with CRS (with/without polyps) and are willing to undergo medical management with antibiotics or steroids, and/or surgical management with functional endoscopic sinus surgery if required

Exclusion Criteria:

* Patients currently having sinonasal tumors - as the middle turbinate may have to be resected in certain cases
* Has undergone functional endoscopic sinus surgery
* Patients with autoimmune diseases affecting the upper airway (e.g. systemic lupus erythematosus, Sjogren's syndrome, systemic sclerosis, etc.)
* Are immuno-compromised, and have impairment in mucociliary function (e.g. cystic fibrosis, Kartagener syndrome)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Modified mini mental state examination | Before starting medical or surgical management and then 6 months after
  This short test consists of questions to assess memory which will take 5-10 minutes to complete.

SECONDARY OUTCOMES:
Change in Cognitive failures Questionnaire | Before starting medical or surgical management and then 6 months after
  This includes 25 questions for patients to self-report everyday errors of perception, memory and motor functioning. It is scored out of 100 with higher score indicating worse more cognitive failures.
Change in Sino-nasal Outcome Test-22 (SNOT-22) scores: | Before starting medical or surgical management and then 6 months after
  This is a standard of care form that includes 22 questions about symptoms and social/emotional consequences of participants nasal disorder. Participants will be asked to rate their problems based on the past two weeks. The questionnaire is out of 110 points with higher score indicating worse symptoms.
Change in Nasal endoscopy | Before starting medical or surgical management and then 6 months after
  This is standard-of-care at St. Paul's Sinus Centre. Participants sinuses will be examined using an instrument called an endoscope which is a metal rod with a camera attached at the end. During the sinus examination, pictures and scores of the sinuses will be recorded. Endoscopic score are given from 0-2 based on endoscopic evidence of polyps, edema and discharge. A higher score indicates worse symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- E.N.T. Clinic, St. Paul's Hospital, Vancouver, British Columbia, Canada